CLINICAL TRIAL: NCT04702997
Title: A Phase 2 Trial to Evaluate Safety, Tolerability, and Efficacy of Bardoxolone Methyl in Patients With Chronic Kidney Disease at Risk of Rapid Progression
Brief Title: A Trial of Bardoxolone Methyl in Patients With CKD at Risk of Rapid Progression (MERLIN)
Acronym: MERLIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 402-C-2002
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Results first posted 2022-12-01 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Chronic Kidney Diseases
Keywords: Advanced CKD; Chronic Kidney Disease; Bardoxolone methyl; RTA 402; eGFR; Advanced Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — bardoxolone methyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bardoxolone methyl (Experimental): Patients randomized to receive bardoxolone methyl capsules orally once daily for 12 weeks at a starting dose of 5 mg and titrated up to a maximal dose of 20 mg (participants with UACR less than or equal to 300 mg/g) or 30 mg (participants with UACR greater than 300 mg/g)
  Patients will be scheduled to be assessed during treatment at Day 1, Weeks 1, 2, 4, 6, 8, and 12 and by telephone contact on Days 3, 10, 21, 31, 35, and 45. Patients will not receive any drug during a 5-week off-treatment period between Weeks 12 and 17. Patients will be assessed on Day 3 off-treatment (OT), Day 7 OT, Day 14 OT, Day 21 OT, Day 28 OT, and Day 35 OT. The OT day corresponds to days after last dose.
  Patients will be assessed at and end-of-study (EOS) visit on Week 17.
  Interventions: Drug: Bardoxolone methyl oral capsule
- Placebo (Placebo Comparator): Patients who received placebo, once-daily, orally, remained on placebo throughout the study duration of 12 weeks and followed the same titration to maintain the blind,
  Patients will be scheduled to be assessed during treatment at Day 1, Weeks 1, 2, 4, 6, 8, and 12 and by telephone contact on Days 3, 10, 21, 31, 35, and 45. Patients will not receive any drug during a 5-week off-treatment period between Weeks 12 and 17. Patients will be assessed on Day 3 off-treatment (OT), Day 7 OT, Day 14 OT, Day 21 OT, Day 28 OT, and Day 35 OT. The OT day corresponds to days after last dose.
  Patients will be assessed at and end-of-study (EOS) visit on Week 17.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Bardoxolone methyl oral capsule — Bardoxolone methyl capsules dose escalated from 5 mg to a maximum of 20 or 30 mg, depending on baseline proteinuria status
  Other Names: RTA 402
  Arms: Bardoxolone methyl
Drug: Placebo oral capsule — Capsule containing an inert placebo
  Arms: Placebo

SUMMARY:
This multi-center, randomized, double-blind, placebo-controlled, Phase 2 trial will study the safety, tolerability, and efficacy of bardoxolone methyl in qualified patients with CKD due to multiple etiologies at risk of rapid disease progression. Approximately 70 patients will be enrolled and randomized 1:1 to either bardoxolone methyl or placebo. Patients with CKD secondary to varying etiologies will be enrolled from age 18-70 years with eGFR ≥ 20 to < 60 mL/min/1.73 m2, and other risk factors for rapid progression of kidney disease.

The maximum target dose will be determined by baseline proteinuria status. Patients with baseline urine albumin to creatinine ratio (UACR) ≤ 300 mg/g will be titrated to a maximum dose of 20 mg, and patients with baseline UACR > 300 mg/g will be titrated to a maximum dose of 30 mg. Qualified patients will be randomized 1:1 to receive either bardoxolone methyl or placebo once daily (preferably in the morning) throughout a 12-week dosing period.

Patients in the study will follow the same visit and assessment schedule. Patients will be assessed during treatment at Day 1, Weeks 1, 2, 4, 6, 8, and 12 and by telephone contact on Days 3, 10, 21, 31, 35, and 45. Date of last dose and the end-of-treatment assessments mark the end of the treatment period. Patients will not receive study drug during a 5-week off-treatment period between Weeks 12 and 17. The off-treatment (OT) period includes 5 visits requiring various assessments to characterize eGFR from the time of study drug discontinuation through Day 35 off-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CKD with screening eGFR (average of Screen A and Screen B eGFR values) ≥ 20 to < 60 mL/min/1.73 m2
* Patient must meet at least one of the following criteria:

  1. UACR ≥ 300 mg/g; OR
  2. eGFR decline at a rate of ≥ 4 mL/min/1.73 m2 in prior year; OR
  3. Hematuria defined as > 5-10 red blood cells (RBCs) per high power field (HPF, manual method), or documented history of positive urinary dipstick for blood in prior year, or macroscopic hematuria in prior 3 years;
* Systolic blood pressure ≤ 150 mmHg and diastolic blood pressure ≤ 90 mmHg at Screen A visit after a period of rest (≥ 5 minutes);
* Treatment with an angiotensin-converting enzyme inhibitor (ACEi) and/or an angiotensin II receptor blocker (ARB) at the maximally tolerated labeled daily dose for at least 6 weeks prior to the Screen A visit and with no anticipated changes to dose(s) during study participation.
* Able to swallow capsules -

Exclusion Criteria:

* Prior exposure to bardoxolone methyl;
* CKD secondary to or associated with any of the following:

  1. History of rapidly progressive glomerulonephritis (RPGN)
  2. Glomerulonephritis requiring immunosuppression in the last 6 months prior to Screen A;
* Concomitant use of tolvaptan.
* Systemic immunosuppression for more than 2 weeks, cumulatively, within the 12 weeks prior to Day 1 or anticipated need for immunosuppression during the study;
* Patients currently taking a sodium/glucose cotransporter-2 inhibitor (SGLT2i), requiring dose adjustments within 12 weeks prior to Day 1 or if dose is anticipated to change during study participation;
* B-type natriuretic peptide (BNP) level > 200 pg/mL at Screen A visit;
* Uncontrolled diabetes (HbA1c > 11.0%) at Screen A visit;
* Serum albumin < 3 g/dL at Screen A visit;
* Kidney or any other solid organ transplant recipient or a planned transplant during the study;
* Acute dialysis or acute kidney injury within 12 weeks prior to Screen A visit or during Screening;
* History of clinically significant cardiac disease;
* Systolic blood pressure < 90 mmHg at Screen A visit after a period of rest;
* Body mass index < 18.5 kg/m2 at the Screen A visit;
* History of malignancy within 5 years prior to Screen A visit, with the exception of localized skin or cervical carcinomas;
* Coronavirus disease 2019 (COVID-19) diagnosis within 3 months prior to Screen A or have ever required COVID-19 related hospitalization;
* Participation in other interventional clinical studies within 3 months (or if relevant 5 half-lives of that study medication, whichever is the longer) prior to Screen B;
* Unwilling to practice acceptable methods of birth control;
* Women who are pregnant or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-11-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - California Institute of Renal Research, La Mesa, California
  - Western Nephrology, Arvada, Colorado
  - Colorado Kidney Care, Denver, Colorado
  - Boise Kidney & Hypertension, PLLC, Nampa, Idaho
  - Renal Associates of Baton Rouge, Baton Rouge, Louisiana
  - Nephrology Center, PC, Kalamazoo, Michigan
  - DaVita Clinical Research, Las Vegas, Nevada
  - Columbia Nephrology Associates, PA, Columbia, South Carolina
  - Renal Disease Research Intitute, Dallas, Texas
  - DaVita Clinical Research, Houston, Texas
  - Gamma Medical Research Inc, McAllen, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Bardoxolone Methyl: Bardoxolone methyl capsules administered orally once daily for 12 weeks at a starting dose of 5 mg and titrated up to a maximal dose of 20 mg (participants with UACR less than or equal to 300 mg/g) or 30 mg (participants with UACR greater than 300 mg/g)
- Placebo: Placebo capsules administered orally once-daily for 12 weeks, with sham titration to maintain the blind.
Period: Overall Study
Arm/Group | Bardoxolone Methyl | Placebo
Started | 39 | 42
Completed | 38 | 41
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo capsules administered orally once daily for 12 weeks, with sham titration to maintain the blind
- Total: Total of all reporting groups
Arm/Group | Bardoxolone Methyl | Placebo | Total
Number analyzed (Participants) | 39 | 42 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (13.5) | 59.8 (12.66) | 58.2 (13.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 23 | 26 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 10 | 27
  Not Hispanic or Latino | 22 | 31 | 53
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 32 | 39 | 71
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 39 | 42 | 81
Baseline estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73 m^2] — eGFR is a measure of kidney function assessed through blood/serum. Higher eGFRs represent better/improved kidney function. Lower eGFRs represent poorer/decreased kidney function.
  mL/min/1.73 m^2 | 36.563 (9.8465) | 34.883 (10.1765) | 35.692 (9.9921)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 12
Description: To assess the change in eGFR from baseline to week 12. eGFR is a measure of kidney function assessed through blood/serum. Higher eGFRs represent better/improved kidney function. Lower eGFRs represent poorer/decreased kidney function.
Time Frame: Baseline through 12 weeks after participant receives the first dose
Population: Intent-to-treat population (all enrolled patients whether or not they received the study drug)
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | Bardoxolone Methyl | Placebo
Number analyzed (Participants) | 39 | 42
mL/min/1.73 m^2 | 6.79 (0.925) | -0.92 (0.868)
Statistical Analysis 1: Comparison: Bardoxolone Methyl vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis — KDIGO strata, treatment group, time (Week 1 to 12), and the interaction between treatment and time were used as fixed factors; LS Mean difference (Net) = 7.71, 95% CI 2-sided [5.18 to 10.24], Standard Error of Mean 1.268 — Difference is bardoxolone methyl - placebo

ADVERSE EVENTS:
Time Frame: 17 weeks
Description: All adverse events that are observed or reported by the patient during the study (from the time of the first dose of study drug until the final visit) must be reported, regardless of their relationship to study drug or their clinical significance.
Arm/Group | Bardoxolone Methyl | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/42
Serious Adverse Events (participants affected / at risk) | 3/39 | 1/42
Other Adverse Events (participants affected / at risk) | 31/39 | 30/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bardoxolone Methyl (N=39) | Placebo (N=42)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bardoxolone Methyl (N=39) | Placebo (N=42)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Cardiac septal hypertrophy (Cardiac disorders) | 1 (1) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 1 (1)
Diabetic retinal oedema (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Macular detachment (Eye disorders) | 1 (1) | 0 (0)
Non-proliferative retinopathy (Eye disorders) | 1 (1) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 6 (8) | 3 (4)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 2 (2)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 2 (3) | 4 (4)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (2)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Corona virus infection (Infections and infestations) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0)
Blood magnesium decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Brain natriuretic peptide increased (Investigations) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 6 (6) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Gout (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Magnesium deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 (9) | 8 (8)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 4 (6)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Meniscus operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT04702997/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT04702997/SAP_001.pdf